CLINICAL TRIAL: NCT03430713
Title: Comparison of Visual and Spectrophotometric Methods for Dental Color Measurement - A Pilot Clinical Trial
Brief Title: Comparison of Visual and Spectrophotometric Methods for Dental Color Measurement - An in Vivo Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Grupo de Investigação em Bioquímica e Biologia Oral (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: I2018-02
Record Dates: First submitted 2018-02-06; First posted 2018-02-13 (Actual); Last update posted 2018-03-02 (Actual); Status verified 2018-03

CONDITIONS: Color Perception; Tooth
Keywords: tooth color; measurement; accuracy; shade guide; spectrophotometer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dental colour measurement (Experimental): Comparison of dental colour measurement between two shade guides VITA Classical and VITA Toothguide 3D-Master and two spectrophotometers VITA Easyshade and Spectroshade Micro
  Interventions: Procedure: Measure of tooth color

INTERVENTIONS:
Procedure: Measure of tooth color — Evaluation of agreement about measure of tooth color between clinicians using two dental shade guides and two spectrophotometers in the determination of the color of maxilary central incisors and canines.

SUMMARY:
Twenty patients of Dental Medicine School will be recruited to participate in a pilot study about dental color measurement in which visual and digital instruments will be tested.

Informed consents and local ethical committee clearance will be previously obtained.

All data will be collected after an oral hygiene procedure. Two different methods of color measurement will be tested: visual method with VITA Classical (VC) and VITA 3D-Master (VM) and digital method with Spectroshade Micro (SS) and VITA Easyshade (ES). The CIE L*a*b* values will be evaluated in the VC scale for both methods. Reproducibility will be assessed based on intra-operator intra-device agreement and the accuracy will be assessed based on inter-device agreement using the kappa coefficient (K) and intraclass correlation coefficient (ICC), respectively. Results will be presented as mean, with 95% CI

DETAILED DESCRIPTION:
Clinical practice in Dentistry has been changed during the times, with a large development of aesthetics considerations.

Tooth color is an effect of volume reflection, the passage of incident light through the tooth followed by backward emergence. Color can be categorized in different systems and CIE L*a*b* is the most common. For color acquision visual and digital methods are used.

Tooth shade matching in daily clinical practice is still a cause of disagreement and discomfort for many professionals. The gold standard is the use of dental shade guides by the clinicans who make a comparison between the sample (tooth) and multiple standard guides (shade guide tabs).

The gold standard visual system has been Vitapan Classical (VC). Other system is Toothguide 3D-Master (VM) which applies more closely the accepted color perception concepts of hue, lightness, chroma.

However, several limitations have been associated to visual procedure. The accuracy between clinicians is frequently low and there is a high variability.

For this reason, many improvements in optical electronic devices have led to the expanded use of photometric and colorimetric techniques for the evaluation, specification and management of color.

Although the effectiveness of these devices depends ultimately on the accuracy and precision with which the measurements are carried out.

There is a deeply concern with the determination of the accuracy between different methods for colour acquision because color has to be communicated precisely.

ELIGIBILITY:
Inclusion Criteria:

* Presence of all upper anterior teeth
* A3 or darker in at least one of those indicated tooth
* Professional dental prophylaxis in last fifteen days

Exclusion Criteria:

* Bleaching treatments in last three years
* Orthodontic appliances in indicated tooth
* Presence of caries
* Color changes
* Dental abnormalities
* Internal spots
* Anterior restorations
* Anterior crowns
* Anterior veneers

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Dental color measurement | 2 weeks
  Agreement between two clinicians using two dental shade guides and two spectrophotometers in the determination of the colour of maxilary central incisors and canines

CONTACTS AND LOCATIONS:
Overall Officials: Duarte Marques, DSD, PhD, Study Director — Grupo de Investigação em Bioquímica e Biologia Oral; Rita Alves, DSD, Principal Investigator — Grupo de Investigação em Bioquímica e Biologia Oral

IPD SHARING:
Plan to Share IPD: No